CLINICAL TRIAL: NCT04792086
Title: The Impact of the COVID-19 Epidemic on the Health of Older Adults
Brief Title: Disease Containment Measures Among Older Adults During the Covid-19 Pandemia
Acronym: Co-AiT
Status: Recruiting | Type: Observational
Sponsor: Norwegian Centre for Ageing and Health (Other)
Responsible Party: Sponsor
Other Study IDs: COVID19-AIT
Record Dates: First submitted 2021-02-02; First posted 2021-03-10 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Dementia; Cognitive Impairment; Depression, Anxiety; Loneliness
Keywords: Dementia; Pandemic; Health care services; Population study; Older adults; Depression
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inhabitants in Nord-Trøndelag 70 years of age and older: All inhabitants in Nord-Trøndelag 70 years of age and older, who participated in the HUNT4 70+-study, between 2017 and 2019.
- Inhabitants in one area in Trondheim, 70 years of age and older: All inhabitants one area in Trondheim, 70 years of age and older, who participated in the HUNT4 70+-study, between 2017 and 2019.

SUMMARY:
This study will examine which impact lockdown strategies intending to prevent the spread of COVID-19 had on people with cognitive impairment and dementia.

Comprehensive data from two large health studies in Norway, conducted before and after the COVID-19 outbreak, will be linked with health register data on the use of health care services and medication. Further, it will be conducted a survey addressing questions on social isolation and use of communicative technology, from March 2020 to January 2021. The knowledge gained from this study can improve the health care system's ability to respond more adequately to pandemics and other unforeseen events, so that the negative consequences for older adults with dementia and cognitive impairment can be reduced.

DETAILED DESCRIPTION:
Introduction: To prevent the spread of COVID-19 societies around the world have implemented various levels of lockdown strategies. Norway locked down major parts of the society from March 2020. Specifically, this meant that public services were closed (e.g. most in-home healthcare services, day care centres, group exercise/gyms and services that offer physiotherapy, medical and psychological consultation). For people with cognitive impairment and dementia, social distancing and self-isolation may have limited the use of normal strategies (e.g., distraction, stimulation, and social interaction) that are routinely adopted to manage some of the dementia symptoms, such as neuropsychiatric symptoms. A lack of daily routines may change the clinical conditions of patients with dementia. Worsening of preexisting and/or the onset of new neuropsychiatric symptoms may occur, in addition to a possible decline of cognitive and functional capacities

Aim: The overarching aim of this project is to provide decision makers with vital information to improve the healthcare of people with dementia and cognitive impairment in the context of an epidemic.

Method: We will use four data sources:1) The fourth wave of the Trøndelag Health study (HUNT, HUNT4 70+), 2) Three national health registries (The Norwegian Patient Registry (NPR), the Norwegian Registry for Primary Health Care (NRPHC) and the Norwegian Prescription Database (NorPD)), 3) A postal questionnaire concerning social isolation during the COVID-19 epidemic, and 4) The Ageing in Trøndelag study (AiT), which is a follow-up of the HUNT4 70+ study.

With this linkage of cohort data and national health registry data, we can identify factors that may make people with cognitive impairment and dementia vulnerable to loss of healthcare services because of COVID-19 and subsequently to negative health consequences.

ELIGIBILITY:
Inclusion Criteria:

* Inhabitants living in the designated areas

Exclusion Criteria:

* None

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Inhabitants living in the designated areas that volunteered to participation in the HUNT4 health survey
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Use of Health care services | The participants' use of health care services from the period 2017-2019
  Information from the Norwegian Patient Registry (NPR) and the Norwegian Registry for Primary Health Care (NRPHC)
Use of Health care services | The participants' use of health care services in 2020
  Information from the Norwegian Patient Registry (NPR) and the Norwegian Registry for Primary Health Care (NRPHC)
Use of Health care services | The participants' use of health care services from the period 2021-2022
  Information from the Norwegian Patient Registry (NPR) and the Norwegian Registry for Primary Health Care (NRPHC)
Use of psychotropic medications | The participants' use of psychotropic medication from the period 2017-2019
  Information from the Norwegian Prescription Database (NorPD)
Use of psychotropic medications | The participants' use of psychotropic medication in 2020
  Information from the Norwegian Prescription Database (NorPD)
Use of psychotropic medications | The participants' use of psychotropic medication from the period 2021-2022
  Information from the Norwegian Prescription Database (NorPD)

SECONDARY OUTCOMES:
Montreal Cognitive Assessment scale | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022
  Tests cognitive function in the domain's memory, visuospatial and executive functions, attention, concentration, language and orientation. Scores from 0 - 30 where 30 indicates best function. impairment or dementia, and questions on subjective memory decline
CERAD Ten-words test | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022
  Tests immediate and delayed memory. Scores from 0 - 30 in immediate memory and 0-10 in delayed recall, higher scores indicates better function.
Incidence of dementia diagnosis | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022
  Two clinical and scientific experts will independently set at diagnosis of cognitive impairment or dementia based on all available information applying standard diagnostic criteria DSM-5
Incidence of mild cognitive impairment | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022
  Two clinical and scientific experts will independently set at diagnosis of cognitive impairment or dementia based on all available information applying standard diagnostic criteria DSM-5

OTHER OUTCOMES:
Short Physical Performance Battery | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022.
  The test combines the results of the gait speed, chair stand and balance test
Grip strength | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022.
  Measured in both hands with a Jamar and digital dynamometer
Blood Pressure | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022
  Systolic blood pressure
Body mass index | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022
  Weight and height will be combined to report BMI in kg/m^2
Upper arm circumference | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022
  The circumference Is measured in centimeters
The Hospital Anxiety and Depression scale | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022
  Gathers information on anxiety and depression, scores from 0 - 42 where 0 indicates best function
Alcohol consumption | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022
  Innhouse made questionnaire about average alcohol units per week and/or month
Physical Self-Maintenance scale | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022
  Assess problems with personal activities of daily living. Assessed in proxy interview and by health personnel for participants in institutions, scores function in 6 personal activities, lower scores indicates better function
Instrumental Activities of daily function | The participants were assessed when attending the HUNT4 70+-study, and will be assessed with the same measures in the followup study in 2021/2022
  Assess problems with instrumental activities of daily living, scores function in 8 instrumental activities, lower scores indicates better function
Social isolation | The participants receive a postal questionnaire in Januar 2021, regarding the period from March 2020-January 20201
  Questions on the experience of social isolation as a result of containment measures due to covid-19, including information on the level of isolation; accepting visits from friends, family or health care services, and restrictions about outdoor activities
Fear of Covid-19 | The participants receive a postal questionnaire in Januar 2021, regarding the period from March 2020-January 20201
  A seven-item scale on fear of covid-19, rated on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree) with scores ranging from 7 to 35. The higher the score, the greater the fear of COVID-19
The use of information and communicative technology (ICT) | The participants receive a postal questionnaire in Januar 2021, regarding the period from March 2020-January 20201
  Questions on the use of ICT, including questions on keeping contact with familly, friend and health care personnel

CONTACTS AND LOCATIONS:
Overall Officials: Geir Selbaek, PhD, Study Director — Norwegian National Advisory Unit on Ageing and Health
Locations (1):
- Norwegian National Advisory Unit of Ageing and Health, Tønsberg, Norway

REFERENCES:
- [Derived] Ibsen TL, Zotcheva E, Bergh S, Gerritsen D, Livingston G, Luras H, Mamelund SE, Rokstad AMM, Strand BH, Voshaar RCO, Selbaek G. Cognitive function, physical function, and mental health in older adults amid reduced primary and specialist healthcare service use during COVID-19: the HUNT study. Geroscience. 2025 Sep 27. doi: 10.1007/s11357-025-01909-x. Online ahead of print. PMID 41006671
- [Derived] Ibsen TL, Zotcheva E, Bergh S, Gerritsen D, Livingston G, Luras H, Mamelund SE, Mork Rokstad AM, Strand BH, Thingstad P, Oude Voshaar RC, Selbaek G. The Role of Social Media in Mitigating the Long-Term Impact of Social Isolation on Mental and Cognitive Health in Older Adults During the COVID-19 Pandemic: The HUNT Study. Int J Geriatr Psychiatry. 2025 May;40(5):e70097. doi: 10.1002/gps.70097. PMID 40338168
- [Derived] Ibsen TL, Zotcheva E, Bergh S, Gerritsen D, Livingston G, Luras H, Mamelund SE, Rokstad AMM, Strand BH, Oude Voshaar RC, Selbaek G. A longitudinal cohort study on dispensed analgesic and psychotropic medications in older adults before, during, and after the COVID-19 pandemic: the HUNT study. BMC Geriatr. 2025 Feb 7;25(1):85. doi: 10.1186/s12877-025-05745-8. PMID 39920618
- [Derived] Ibsen TL, Strand BH, Bergh S, Livingston G, Luras H, Mamelund SE, Voshaar RO, Rokstad AMM, Thingstad P, Gerritsen D, Selbaek G. A longitudinal cohort study on the use of health and care services by older adults living at home with/without dementia before and during the COVID-19 pandemic: the HUNT study. BMC Health Serv Res. 2024 Apr 19;24(1):485. doi: 10.1186/s12913-024-10846-y. PMID 38641570